CLINICAL TRIAL: NCT04485416
Title: Open Label Single Arm Prospective Pilot Trial of Eltrombopag in Patients 1 Year to 18 Years of Age Undergoing Intensive Chemotherapy for Malignant Solid Tumors (CCPO011)
Brief Title: Pilot Trial of Eltrombopag in Patients Undergoing Chemotherapy for Malignant Solid Tumors
Acronym: CCPO011
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: PI discretion; suspended while CAPA is reviewed
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1602666; 150124 (Other: FDA (IND)); CCPO011 (Other: UC Davis Comprehensive Cancer Center)
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor, Childhood; Solid Tumor
Keywords: chemotherapy; pediatric
MeSH Terms: interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Subjects will receive eltrombopag
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag is an orally administered small-molecule nonpeptide TPO-R agonist.
  Other Names: Promacta

SUMMARY:
Primary Objective: To assess safety of eltrombopag in pediatric patients undergoing intensive chemotherapy for malignant solid tumors.

Secondary Objectives: To assess the efficacy of eltrombopag in increasing platelet count up to 2 weeks after completion of chemotherapy in pediatric patients undergoing intensive chemotherapy for malignant solid tumors.

Hypothesis: The hypothesis is that eltrombopag an oral thrombopoietin receptor agonist will increase the platelet count safely and efficaciously in children having chemotherapy induced thrombocytopenia while on therapy for solid tumors.

DETAILED DESCRIPTION:
Eltrombopag is an orally administered, small molecule thrombopoietin receptor (TPO-R) agonist that stimulates platelet production by a mechanism similar, but not identical to endogenous TPO. Eltrombopag interacts with the transmembrane domain of the TPO-R (also known as C-MPL) leading to increased platelet production (Erickson-Miller, 2010; Sun et al, 2012).

Eltrombopag is indicated for the treatment of thrombocytopenia in adult and pediatric patients one year and older with chronic immune (idiopathic) thrombocytopenia (ITP) who have had an insufficient response to corticosteroids, immunoglobulins, or splenectomy.

Eltrombopag has also been approved for the treatment of thrombocytopenia in adult patients with chronic hepatitis C to allow for the initiation and maintenance of interferon-based therapy and for the treatment of cytopenias in adult patients with severe aplastic anemia (SAA) who have had insufficient responses to immunosuppressive therapy.

This is an open label, single center pilot trial of eltrombopag in pediatric patients receiving cancer directed therapy for solid tumors. The purpose of this study is to explore the platelet supportive care effects and safety of eltrombopag in pediatric patients (ages one to 18 years of age) undergoing intensive chemotherapy for malignant solid tumors. The primary endpoint will be to determine the safety of eltrombopag in pediatric patients undergoing intensive chemotherapy for malignant solid tumors using CTCAE v5.0 criteria. The secondary endpoint will be to determine the efficacy of eltrombopag in pediatric patients undergoing intensive chemotherapy for malignant solid tumors. These objectives will be assessed by evaluating drug-related toxicities, the platelet response in patients and the proportion of subjects receiving eltrombopag who are platelet transfusion-free during the time period of chemotherapy.

The study will enroll 10 subjects with histologically confirmed solid tumors, including but not limited to rhabdomyosarcoma, Ewing sarcoma, osteosarcoma, non-rhabdomyosarcoma soft tissue sarcoma, peripheral nerve sheath tumor, desmoplastic small round cell tumor, hepatoblastoma, hepatocellular carcinoma, renal cell carcinoma, higher grade neuroblastoma, medulloblastoma, or other rare malignant solid tumors.

The cancer directed therapy will be part of standard treatment for each patient and will consist of two to four cycles of chemotherapy (or as many as clinically indicated per physician discretion) to reduce tumor burden, followed by surgery in the majority of cases, and/or radiation in a minority of cases, or both in rare cases at various times in the course of treatment. After recovery from the surgery and/or radiation, chemotherapy and eltrombopag will be resumed until completion. Each cycle of chemotherapy will be approximately two to four weeks (14 to 28 days) in length with chemotherapy administered for one to five days per cycle. The duration of chemotherapy varies by regimen and underlying malignancy.

Patients will initiate eltrombopag on the first day following the completion of chemotherapy for each cycle (e.g., chemo is administered on Days 1-5, eltrombopag to start on Day 6). Eltrombopag will be administered daily and the dose will be age dependent (see Table 5). Children less than 6 years of age will receive a starting dose of 25 mg by mouth once daily, taken on empty stomach one hour before or two hours after a meal. For children greater than or equal to 6 years of age, the starting dose will be 75 mg by mouth once daily. Doses shall be reduced in patients of Asian ancestry (e.g., Japanese, Chinese, Taiwanese, or Korean): for those patients greater than or equal to 6 years of age, the starting dose will be 50 mg by mouth once daily and for those patients less than 6 years old, the starting dose will be 12.5 mg by mouth once daily. Eltrombopag will be continued until the platelets are at least 100,000/µL after the nadir.

Subjects will be recruited from the UC Davis Comprehensive Cancer Center or when they are admitted to UC Davis Children's Hospital.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for study entry.

1. Persons aged ≥ 1 to ≤18 years of age.
2. Histologically confirmed solid tumors (including rhabdomyosarcoma, Ewings sarcoma, osteosarcoma, non- rhabdomyosarcoma soft tissue sarcoma, peripheral nerve sheath tumor, desmoplastic small round cell tumor, hepatoblastoma, hepatocellular carcinoma, renal cell carcinoma, higher grade neuroblastoma, brain tumors (e.g. medulloblastoma), and other rare solid tumors.
3. Currently receiving cancer directed therapy for solid tumor or scheduled to start receiving cancer directed therapy for solid tumor within 60 days.
4. Karnofsky Performance Status (KPS) performance status of 80% or greater.
5. Life expectancy ≥ 6 months.
6. Ability to swallow liquid solution/suspensions or tablets/capsules
7. Platelet count < 150,000µL
8. Blood chemistry levels defined by:

   * Serum creatinine less than or equal to 2.5 × the upper limit of normal (ULN) range
   * Total bilirubin level less than or equal to 1.5 × the upper limit of normal (ULN) range
   * AST and ALT < 3 x upper limit of normal (ULN)
9. INR and aPTT less than or equal to 1.5 × ULN (for patients on anticoagulation they must be receiving a stable dose for at least 1 week prior to first treatment)
10. Ability to understand and willingness to sign an informed consent form; or Parent/Guardian with ability to understand and willingness to sign an informed consent form.
11. Ability to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry.

1. Patients with known with hematologic malignancy diagnosis.
2. Contraindications to receiving chemotherapy.
3. Patients with history of thromboembolic disease or history of thrombophilic risk factors.
4. History or current diagnosis of cardiac disease indicating significant risk of safety for patients participating in the study such as uncontrolled or significant cardiac disease, including any of the following:

   * Recent myocardial infarction (within last 6 months),
   * Uncontrolled congestive heart failure,
   * Unstable angina (within last 6 months),
   * Clinically significant (symptomatic) cardiac arrhythmias (e.g., sustained ventricular tachycardia, and clinically significant second or third degree AV block without a pacemaker.)
   * Long QT syndrome, family history of idiopathic sudden death, congenital long QT syndrome or additional risk factors for cardiac repolarization abnormality, as determined by the investigator.
5. Impaired cardiac function, defined as:

   * Corrected QTc >450 msec using Fridericia correction (QTcF) on the screening ECG (using triplicate ECGs),
   * Other clinically significant cardio-vascular disease (e.g., uncontrolled hypertension, history of labile hypertension),
   * History of known structural abnormalities (e.g. cardiomyopathy).
6. Pregnant or lactating women.
7. Subjects with liver enzymes 5x upper limit of normal or liver cirrhosis (as determined by the investigator).
8. Patients with known history of HIV positivity.
9. Patient with known active or uncontrolled infections not responding to appropriate therapy.
10. History of alcohol/drug abuse.
11. Concurrent participation in an investigational study within 30 days prior to enrollment or within 8 days (> than 5-half-lives)of the investigational product, whichever is longer. Note: parallel enrollment in a disease registry is permitted.
12. Known thrombophilic risk factors or history of thromboembolic disease. Exception: Subjects for whom the potential benefits of participating in the study outweigh the potential risks of thromboembolic events, as determined by the investigator.
13. Known immediate or delayed hypersensitivity reaction to eltrombopag or its excipient.
14. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using basic methods of contraception during dosing of study treatment. Basic contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening). The vasectomized male partner should be the sole partner for that subject.
    * Barrier methods of contraception: Condom or Occlusive cap.
    * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception. In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
15. Female subjects who are nursing or pregnant (positive serum or urine B-human chorionic gonadotrophin (B-hCG) pregnancy test) at screening or pre-dose on Day 1.
16. Sexually active males unless they use a condom during intercourse while taking the drug during treatment, and for 8 days (> 5 half-lives ) after stopping eltrombopag and for 5 half-lives after the last dose of chemotherapy treatment and should not father a child in this period. A condom is required to be used also by vasectomized men as well as during intercourse with a male partner in order to prevent delivery of the drug via semen.
17. Any condition that would prohibit the understanding or rendering of informed consent.
18. Any condition that in the opinion of the investigator would interfere with the patient's safety or compliance on trial.
19. Severe infection within 4 weeks prior to enrollment that in the opinion of the investigator would interfere with patient safety or compliance on trial.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-07-16 (Actual); Primary Completion 2025-05-17 (Estimated); Study Completion 2025-05-17 (Estimated)

PRIMARY OUTCOMES:
Safety objectives | Through follow up after end of treatment
  For safety our end point is liver enzymes ALT, AST up to 5 x upper limit of normal (ULN) in <80% of patients.

SECONDARY OUTCOMES:
Efficacy objectives | 2 weeks after completion of chemotherapy
  For efficacy the end point is 6 of 10 patients respond to the study treatment by an increase in platelet counts by 20,000/μL and are able to proceed with their next cycle of chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Pawar, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Health System, Comprehensive Cancer Center, Sacramento, California, United States

REFERENCES:
- [Background] Geng W, Kearney S, Nelson S. Upfront eltrombopag monotherapy induces stable hematologic remission in pediatric patients with nonsevere idiopathic aplastic anemia. Pediatr Blood Cancer. 2018 Oct;65(10):e27290. doi: 10.1002/pbc.27290. Epub 2018 Jun 22. PMID 29932285
- [Background] Townsley DM, Scheinberg P, Winkler T, Desmond R, Dumitriu B, Rios O, Weinstein B, Valdez J, Lotter J, Feng X, Desierto M, Leuva H, Bevans M, Wu C, Larochelle A, Calvo KR, Dunbar CE, Young NS. Eltrombopag Added to Standard Immunosuppression for Aplastic Anemia. N Engl J Med. 2017 Apr 20;376(16):1540-1550. doi: 10.1056/NEJMoa1613878. PMID 28423296
- [Background] Soff GA, Miao Y, Bendheim G, Batista J, Mones JV, Parameswaran R, Wilkins CR, Devlin SM, Abou-Alfa GK, Cercek A, Kemeny NE, Sarasohn DM, Mantha S. Romiplostim Treatment of Chemotherapy-Induced Thrombocytopenia. J Clin Oncol. 2019 Nov 1;37(31):2892-2898. doi: 10.1200/JCO.18.01931. Epub 2019 Sep 23. PMID 31545663
- [Background] Li S, Wu R, Wang B, Fu L, Zhu G, Zhou X, Ma J, Zhang L, Qin M. Eltrombopag for Delayed Platelet Recovery and Secondary Thrombocytopenia Following Allogeneic Stem Cell Transplantation in Children. J Pediatr Hematol Oncol. 2019 Jan;41(1):38-41. doi: 10.1097/MPH.0000000000001263. PMID 30080752
- [Background] Erickson-Miller CL, Kirchner J, Aivado M, May R, Payne P, Chadderton A. Reduced proliferation of non-megakaryocytic acute myelogenous leukemia and other leukemia and lymphoma cell lines in response to eltrombopag. Leuk Res. 2010 Sep;34(9):1224-31. doi: 10.1016/j.leukres.2010.02.005. Epub 2010 Mar 3. PMID 20202683
- [Background] Sun H, Tsai Y, Nowak I, Liesveld J, Chen Y. Eltrombopag, a thrombopoietin receptor agonist, enhances human umbilical cord blood hematopoietic stem/primitive progenitor cell expansion and promotes multi-lineage hematopoiesis. Stem Cell Res. 2012 Sep;9(2):77-86. doi: 10.1016/j.scr.2012.05.001. Epub 2012 May 14. PMID 22683680
- [Background] Ballmaier M, Germeshausen M, Krukemeier S, Welte K. Thrombopoietin is essential for the maintenance of normal hematopoiesis in humans: development of aplastic anemia in patients with congenital amegakaryocytic thrombocytopenia. Ann N Y Acad Sci. 2003 May;996:17-25. doi: 10.1111/j.1749-6632.2003.tb03228.x. PMID 12799278
- [Background] Zeigler FC, de Sauvage F, Widmer HR, Keller GA, Donahue C, Schreiber RD, Malloy B, Hass P, Eaton D, Matthews W. In vitro megakaryocytopoietic and thrombopoietic activity of c-mpl ligand (TPO) on purified murine hematopoietic stem cells. Blood. 1994 Dec 15;84(12):4045-52. PMID 7527664
- [Background] Qian H, Buza-Vidas N, Hyland CD, Jensen CT, Antonchuk J, Mansson R, Thoren LA, Ekblom M, Alexander WS, Jacobsen SE. Critical role of thrombopoietin in maintaining adult quiescent hematopoietic stem cells. Cell Stem Cell. 2007 Dec 13;1(6):671-84. doi: 10.1016/j.stem.2007.10.008. Epub 2007 Nov 20. PMID 18371408
- [Background] Erickson-Miller CL, Delorme E, Tian SS, Hopson CB, Landis AJ, Valoret EI, Sellers TS, Rosen J, Miller SG, Luengo JI, Duffy KJ, Jenkins JM. Preclinical activity of eltrombopag (SB-497115), an oral, nonpeptide thrombopoietin receptor agonist. Stem Cells. 2009 Feb;27(2):424-30. doi: 10.1634/stemcells.2008-0366. PMID 19038790
- [Background] Alexander WS, Roberts AW, Nicola NA, Li R, Metcalf D. Deficiencies in progenitor cells of multiple hematopoietic lineages and defective megakaryocytopoiesis in mice lacking the thrombopoietic receptor c-Mpl. Blood. 1996 Mar 15;87(6):2162-70. PMID 8630375
- [Background] Kimura S, Roberts AW, Metcalf D, Alexander WS. Hematopoietic stem cell deficiencies in mice lacking c-Mpl, the receptor for thrombopoietin. Proc Natl Acad Sci U S A. 1998 Feb 3;95(3):1195-200. doi: 10.1073/pnas.95.3.1195. PMID 9448308
- [Background] Kellum A, Jagiello-Gruszfeld A, Bondarenko IN, Patwardhan R, Messam C, Mostafa Kamel Y. A randomized, double-blind, placebo-controlled, dose ranging study to assess the efficacy and safety of eltrombopag in patients receiving carboplatin/paclitaxel for advanced solid tumors. Curr Med Res Opin. 2010 Oct;26(10):2339-46. doi: 10.1185/03007995.2010.510051. PMID 20735290
- [Background] Olnes MJ, Scheinberg P, Calvo KR, Desmond R, Tang Y, Dumitriu B, Parikh AR, Soto S, Biancotto A, Feng X, Lozier J, Wu CO, Young NS, Dunbar CE. Eltrombopag and improved hematopoiesis in refractory aplastic anemia. N Engl J Med. 2012 Jul 5;367(1):11-9. doi: 10.1056/NEJMoa1200931. PMID 22762314